CLINICAL TRIAL: NCT00414986
Title: Using Learning Teams for Reflective Adaptation
Brief Title: Using Learning Teams for Reflective Adaptation for Diabetes and Depression
Acronym: ULTRA-DM/MDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 05-0457; R18DK067083 (NIH); MH069806
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Type 2 Diabetes; Hyperlipidemia; Hypertension; Depression
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperlipidemias; Hypertension; Depression | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Practice in this arm will receive the Chronic Care Improvement intervention
  Interventions: Behavioral: Chronic Care Improvement (CCI) Intervention
- 2 (Experimental): Practices in this arm will receive the standard CQI intervention. An in-practice CQI coordinator will assist the practices in implement a chronic disease registry.
  Interventions: Behavioral: Standard CQI intervention
- 3 (Active Comparator): Practice in this arm will have access to all chronic care tools, but will not have an in-practice change agent.
  Interventions: Behavioral: Self-directed practice comparison

INTERVENTIONS:
Behavioral: Standard CQI intervention — In-practice change facilitator assists the practice in implementing a chronic disease registry
  Arms: 2
Behavioral: Chronic Care Improvement (CCI) Intervention — An in-practice change facilitator will assist the Improvement Team in enhancing the relationship infrastructure of the practice and in implementing diabetes and depression office systems.
  Arms: 1
Behavioral: Self-directed practice comparison — Practices will have access to all tools used in Arm 1 via a project website
  Arms: 3

SUMMARY:
The study will randomize 54 primary care practices to two intervention and a comparison groups. Both interventions will involve an on-site Improvement Facilitator who will assist the practice in forming an Improvement Team, using rapid-cycle tests of change, and implementing chronic care office systems for type 2 diabetes and depression. One intervention is based on complexity science and the other is a traditional QI intervention.

DETAILED DESCRIPTION:
Evidence-based guidelines for primary care of diabetes have been established and disseminated, yet adoption of guidelines in community-based primary care practice has been disappointing. This effectiveness study proposes a randomized trial involving 54 community-based primary care practices to test two innovative interventions to improve diabetes and depression care. One intervention, derived from theoretically based and efficacious programs tested in other settings, adopts a broad focus and seeks to improve diabetes and depression care by a) increasing the practice's organizational capacity to manage change, and b) implementing and sustaining chronic care office systems that support clinician efforts to improve care for diabetes. The intervention will combine two integrated components. The first component will utilize an Improvement Facilitator that will assess the practice's current use of chronic care office systems and their organizational capacity to manage change, provide feedback to key stakeholders in the practice, and work with the practice over six months to form an Improvement Team that will both address organizational capacity to create and sustain improvement and implement chronic care systems. In the second component of the intervention, the practice will participate in a local Improvement Collaborative that will afford opportunities to learn and share experiences during implementation and maintenance phases of the intervention with five similar practices in their geographic area. The second intervention is based on traditional QI methods and focuses on a chronic disease registry with regular reports to the physicians. It also uses PDSA cycles to assist in implementing change. This intervention will offer tools to improve diabetes and/or asthma care. Both interventions will be evaluated in two ways. First, a randomized trial using rigorous quantitative methods will measure 2 primary and 3 secondary endpoints at 9 and 18 months, including a) the ADA Physician Recognition Program performance measures by both patient-report and review of the medical record, and b) HEDIS measures of acute phase management of depression, c) assessment of the extent to which practices implement and physicians use elements of the chronic care model in their care of diabetes and depression. Change from baseline to 9 months will assess adoption of chronic care improvements, and change from 9 to 18 months will assess sustainability of improvements. Second, a multimethod assessment process will be used to analyze all qualitative and quantitative data separately to understand how and why the intervention led to the observed effects. The practice assessment will strive to understand which components of the interventions were most effective, their relative costs for implementation, and how they might be further improved. Successful components of the intervention will be refined and made available to our collaborators in the project; the Copic Insurance Company and the Colorado Clinical Guidelines Collaborative, for use in their statewide activities to improve diabetes care.

ELIGIBILITY:
Inclusion Criteria:

* Under primary care for type 2 diabetes

Exclusion Criteria:

* Are not minimally literate in either English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1565 (Actual)
Dates: Start 2005-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Surveillance of Hemoglobin A1c, blood pressure, lipids, depression process of care | Baseline, 9, and 18 month
HEDIS-like measures of acute phase management of depression | Baseline, 9, and 18 months

SECONDARY OUTCOMES:
Patient report (by survey) of their primary care experience | baseline, 9-months, 18-months

CONTACTS AND LOCATIONS:
Overall Officials: David West, PhD, Principal Investigator — Department of Family Medicine, University of Colorado Health Sciences Center
Locations (1):
- University of Colorado Health Sciences Center, Denver, Colorado, United States